CLINICAL TRIAL: NCT06903260
Title: Robot-assisted Partial Nephrectomy With and Without Mixed Reality (REALITATEM Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Brainlab AG (Industry); Magic Leap Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66791623.8.0000.5330
Record Dates: First submitted 2025-02-26; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Kidney Cancer
Keywords: Robot-assisted Partial Nephrectomy; Mixed Reality; Augmented Reality; Virtual Reality; Ischemia Time
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient's accrual occurred in the private clinic of a few urologists, and patients were blinded to the intervention they would be submitted to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Realitatem Group (Experimental): robot assisted partial nephrectomy with use of mixed reality
  Interventions: Combination Product: Mixed Reality
- Control group (No Intervention): robot assisted partial nephrectomy with out use of mixed reality

INTERVENTIONS:
Combination Product: Mixed Reality — Virtual reality (VR) is defined as an artificial 3D visual environment and augmented reality (AR), as virtual objects superimposed on the real world; mixed reality is the association between VR and AR. The images were exported from CT image in DICOM (Digital Imaging and Communications in Medicine) and applied in Brainlab Elements software (Brainlab AG, Munich, Germany), where the images and 3D drawing were rendered in partnership with the collaborating bioengineer of this work to obtain the VR. AG was obtained during the intraoperative through the Magic Leap 1 goggle (Magic Leap Inc., Plantation, FL, USA)
  Arms: Realitatem Group

SUMMARY:
Kidney cancer has had a raising diagnostic incidence and partial nephrectomy (PN) is the standard of care for renal masses stage cT1a and a possible treatment choice for cT1b/T2; PN may be associated to a variety of tools, such as three-dimensional (3D) models, which can be used as printed models or through VR (virtual reality) and/or AR (augmented reality). Virtual reality is defined as an artificial 3D visual environment and AR, as virtual objects superimposed on the real world; mixed reality (MIXREAL) is the association between VR and AR.

The first clinical experience using AR in a PN was in 2008, and since then, clinical trials of 3D assisted minimally invasive PN have been developed, such as the first trial evaluating both AR and VR in videolaparoscopic PN, a prospective cohort, and the first randomized clinical trial evaluating 3D model in robot assisted PN (RAPN), but using only VR; posteriorly, Porpiglia et al. and Li et al. published clinical trials of RAPN using AR.

The investigators aimed to establish the improvements that use of MIXREAL can provide in perioperatory and functional outcomes of RAPN. Although previous studies have been showing positive results on behalf of 3D virtual models, besides this being the first study in Latin America to employ MIXREAL in minimally invasive PN, it is the first randomized clinical trial to employ both AR and VR in the context of RAPN.

To analyze the efficacy of MIXREAL, the investigators intended to allocate forty-five patients with renal lesions to RAPN with, Realitatem Group (RG), or without, Control Group (CG), use of MIXREAL.

DETAILED DESCRIPTION:
Kidney cancer has had a raising diagnostic incidence and partial nephrectomy (PN) is the standard of care for renal masses stage cT1a and a possible treatment choice for cT1b/T2; PN may be associated to a variety of tools, such as three-dimensional (3D) models, which can be used as printed models or through VR (virtual reality) and/or AR (augmented reality). Virtual reality is defined as an artificial 3D visual environment and AR, as virtual objects superimposed on the real world; mixed reality (MIXREAL) is the association between VR and AR.

The first clinical experience using AR in a PN was in 2008, and since then, clinical trials of 3D assisted minimally invasive PN have been developed, such as the first trial evaluating both AR and VR in videolaparoscopic PN, a prospective cohort, and the first randomized clinical trial evaluating 3D model in robot assisted PN (RAPN), but using only VR; posteriorly, Porpiglia et al. and Li et al. published clinical trials of RAPN using AR.

The investigators aimed to establish the improvements that use of MIXREAL can provide in perioperatory and functional outcomes of RAPN. Although previous studies have been showing positive results on behalf of 3D virtual models, besides this being the first study in Latin America to employ MIXREAL in minimally invasive PN, it is the first randomized clinical trial to employ both AR and VR in the context of RAPN.

To analyze the efficacy of MIXREAL, the investigators intended to allocate forty-five patients with renal lesions to RAPN with, Realitatem Group (RG), or without, Control Group (CG), use of MIXREAL.

Patient's accrual occurred in the private clinic of a few urologists, and patients were blinded to the intervention they would be submitted to. The randomization process was done in a manual pattern, where the next case would always be enrolled to a different group than the previous, starting the study with a patient enrolled to RG.

Besides sociodemographic data, pre-operative data regarding the tumor also was collected and it was determined by an updated CT, done within one month from the surgery. Patients randomized to RG were specifically required an angioCT. The images were exported in DICOM (Digital Imaging and Communications in Medicine) and applied in Brainlab Elements software (Brainlab AG, Munich, Germany), where the images and 3D drawing were rendered in partnership with the collaborating bioengineer of this work to obtain the VR (Figure 1). Planned cases were available via cloud services for immediate use in the operating room (www.brainlab.com).

All surgeries were robot-assisted, conducted transperitoneally, and executed at Moinhos de Vento Hospital (Porto Alegre, Rio Grande do Sul), a tertiary center, from August 2022 to January 2024 by 8 urologists with experience in RAPN. AG was obtained through the Magic Leap 1 goggle (Magic Leap Inc., Plantation, FL, USA) (Figure 5); the only role Brainlab and Magic Leap industries had in this study was the providing of the software and the goggle free of charge.

Besides tumor and patient's baseline characteristics and intra-operative data, such as vessel clamping, ischemia time, estimated blood loss (EBL), use of hemostatic agents and excision technique, post-operative data, such as renal function, anatomopathology, complication rate and hospital staying, were also recorded. Our primary endpoint was ischemia time and the rest were secondary endpoints.

The results obtained were stored in a confidential database, with exclusive access to the researchers, and later organized in the Statistical Package for the Social Sciences (SPSS), proceeding to statistical analyzes.

Initially, descriptive analyzes were performed to characterize the sample of participants. Later, comparisons were made between GR and GC through non-parametric tests Mann-Whitney, Chi-square (CH2) and, when necessary, Fisher's exact test. These comparisons constituted homogeneity analyzes between the groups in the case of sociodemographic, preoperative and histopathological characteristics, while in the perioperative and functional variables they served to find a possible difference related to whether or not to use MIXREAL. For all analyzes performed, it was adopted the 95% confidence interval and the significance level of 5% (p ≤ .05).

The sample was calculated using the Risk Calc software. Assuming a difference in mean ischemia rate (primary outcome) between treatment groups to be 3.9 minutes (20), an expected population standard deviation to be 3.23 (11) and a clinically relevant difference to be of 1 minute (22), to achieve 80% power (i.e., 1-β=0.8) at the level of significance of 5% (α=0.05) with equal allocation (i.e., k=1) and dropout rate of 5%, a total sample of at least 34 patients, divided into two groups, would be required

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years old with solid renal masses or complex renal cysts Bosniak III/IV requiring partial nephrectomy

Exclusion Criteria:

* solid renal masses or complex renal cysts Bosniak III/IV with initial indication of radical nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
ischemia time | "Perioperative/Periprocedural"
  time from renal artery clamping to its disclamping

SECONDARY OUTCOMES:
total surgical time | "Perioperative/Periprocedural"
  from first skin incision to skin suture
conversion to open surgery | "Perioperative/Periprocedural"
  conversion to open surgery
artery clamping | "Perioperative/Periprocedural"
  need of artery clamping or off clamp
selective clamping | "Perioperative/Periprocedural"
  clamping of a renal artery branch, instead of the main renal artery
estimated blood loss | "Perioperative/Periprocedural"
  in ml
excision technique | "Perioperative/Periprocedural"
  Wedge resection or Enucleoresection or Enucleation
conversion to radical nephrectomy | "Perioperative/Periprocedural"
  yes or no
perioperative complication | Up to 4 weeks
  according to clavien-dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Andre Kives Berger, MSc, Study Chair — Hospital Moinhos de Vento
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Brazil

REFERENCES:
- [Result] Palumbo C, Pecoraro A, Knipper S, Rosiello G, Luzzago S, Deuker M, Tian Z, Shariat SF, Simeone C, Briganti A, Saad F, Berruti A, Antonelli A, Karakiewicz PI. Contemporary Age-adjusted Incidence and Mortality Rates of Renal Cell Carcinoma: Analysis According to Gender, Race, Stage, Grade, and Histology. Eur Urol Focus. 2021 May;7(3):644-652. doi: 10.1016/j.euf.2020.05.003. Epub 2020 May 23. PMID 32456993
- [Result] Bukavina L, Bensalah K, Bray F, Carlo M, Challacombe B, Karam JA, Kassouf W, Mitchell T, Montironi R, O'Brien T, Panebianco V, Scelo G, Shuch B, van Poppel H, Blosser CD, Psutka SP. Epidemiology of Renal Cell Carcinoma: 2022 Update. Eur Urol. 2022 Nov;82(5):529-542. doi: 10.1016/j.eururo.2022.08.019. Epub 2022 Sep 10. PMID 36100483
- [Result] Motzer RJ, Jonasch E, Boyle S, Carlo MI, Manley B, Agarwal N, Alva A, Beckermann K, Choueiri TK, Costello BA, Derweesh IH, Desai A, George S, Gore JL, Haas N, Hancock SL, Kyriakopoulos C, Lam ET, Lau C, Lewis B, Madoff DC, McCreery B, Michaelson MD, Mortazavi A, Nandagopal L, Pierorazio PM, Plimack ER, Ponsky L, Ramalingam S, Shuch B, Smith ZL, Somer B, Sosman J, Dwyer MA, Motter AD. NCCN Guidelines Insights: Kidney Cancer, Version 1.2021. J Natl Compr Canc Netw. 2020 Sep;18(9):1160-1170. doi: 10.6004/jnccn.2020.0043. PMID 32886895
- [Result] Wake N, Nussbaum JE, Elias MI, Nikas CV, Bjurlin MA. 3D Printing, Augmented Reality, and Virtual Reality for the Assessment and Management of Kidney and Prostate Cancer: A Systematic Review. Urology. 2020 Sep;143:20-32. doi: 10.1016/j.urology.2020.03.066. Epub 2020 Jun 12. PMID 32535076
- [Result] Detmer FJ, Hettig J, Schindele D, Schostak M, Hansen C. Virtual and Augmented Reality Systems for Renal Interventions: A Systematic Review. IEEE Rev Biomed Eng. 2017;10:78-94. doi: 10.1109/RBME.2017.2749527. Epub 2017 Sep 6. PMID 28885161
- [Result] Ukimura O, Gill IS. Imaging-assisted endoscopic surgery: Cleveland Clinic experience. J Endourol. 2008 Apr;22(4):803-10. doi: 10.1089/end.2007.9823. PMID 18366316
- [Result] Wang D, Zhang B, Yuan X, Zhang X, Liu C. Preoperative planning and real-time assisted navigation by three-dimensional individual digital model in partial nephrectomy with three-dimensional laparoscopic system. Int J Comput Assist Radiol Surg. 2015 Sep;10(9):1461-8. doi: 10.1007/s11548-015-1148-7. Epub 2015 Jan 11. PMID 25577366
- [Result] Shirk JD, Thiel DD, Wallen EM, Linehan JM, White WM, Badani KK, Porter JR. Effect of 3-Dimensional Virtual Reality Models for Surgical Planning of Robotic-Assisted Partial Nephrectomy on Surgical Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911598. doi: 10.1001/jamanetworkopen.2019.11598. PMID 31532520
- [Result] Porpiglia F, Checcucci E, Amparore D, Piramide F, Volpi G, Granato S, Verri P, Manfredi M, Bellin A, Piazzolla P, Autorino R, Morra I, Fiori C, Mottrie A. Three-dimensional Augmented Reality Robot-assisted Partial Nephrectomy in Case of Complex Tumours (PADUA >/=10): A New Intraoperative Tool Overcoming the Ultrasound Guidance. Eur Urol. 2020 Aug;78(2):229-238. doi: 10.1016/j.eururo.2019.11.024. Epub 2019 Dec 30. PMID 31898992
- [Result] Li L, Zeng X, Yang C, Un W, Hu Z. Three-dimensional (3D) reconstruction and navigation in robotic-assisted partial nephrectomy (RAPN) for renal masses in the solitary kidney: A comparative study. Int J Med Robot. 2022 Feb;18(1):e2337. doi: 10.1002/rcs.2337. Epub 2021 Oct 10. PMID 34591353
- [Result] Yoshida S, Sugimoto M, Fukuda S, Taniguchi N, Saito K, Fujii Y. Mixed reality computed tomography-based surgical planning for partial nephrectomy using a head-mounted holographic computer. Int J Urol. 2019 Jun;26(6):681-682. doi: 10.1111/iju.13954. Epub 2019 Mar 25. No abstract available. PMID 30912180
- [Result] Edgcumbe P, Singla R, Pratt P, Schneider C, Nguan C, Rohling R. Follow the light: projector-based augmented reality intracorporeal system for laparoscopic surgery. J Med Imaging (Bellingham). 2018 Apr;5(2):021216. doi: 10.1117/1.JMI.5.2.021216. Epub 2018 Feb 14. PMID 29487888
- [Result] Porpiglia F, Fiori C, Checcucci E, Amparore D, Bertolo R. Hyperaccuracy Three-dimensional Reconstruction Is Able to Maximize the Efficacy of Selective Clamping During Robot-assisted Partial Nephrectomy for Complex Renal Masses. Eur Urol. 2018 Nov;74(5):651-660. doi: 10.1016/j.eururo.2017.12.027. Epub 2018 Jan 6. PMID 29317081
- [Result] Scosyrev E, Messing EM, Sylvester R, Campbell S, Van Poppel H. Renal function after nephron-sparing surgery versus radical nephrectomy: results from EORTC randomized trial 30904. Eur Urol. 2014 Feb;65(2):372-7. doi: 10.1016/j.eururo.2013.06.044. Epub 2013 Jul 2. PMID 23850254
- [Result] Alrumayyan M, Raveendran L, Lawson KA, Finelli A. Cystic Renal Masses: Old and New Paradigms. Urol Clin North Am. 2023 May;50(2):227-238. doi: 10.1016/j.ucl.2023.01.003. Epub 2023 Feb 20. PMID 36948669
- [Result] Moch H, Amin MB, Berney DM, Comperat EM, Gill AJ, Hartmann A, Menon S, Raspollini MR, Rubin MA, Srigley JR, Hoon Tan P, Tickoo SK, Tsuzuki T, Turajlic S, Cree I, Netto GJ. The 2022 World Health Organization Classification of Tumours of the Urinary System and Male Genital Organs-Part A: Renal, Penile, and Testicular Tumours. Eur Urol. 2022 Nov;82(5):458-468. doi: 10.1016/j.eururo.2022.06.016. Epub 2022 Jul 16. PMID 35853783
- [Result] Ljungberg B, Hanbury DC, Kuczyk MA, Merseburger AS, Mulders PF, Patard JJ, Sinescu IC; European Association of Urology Guideline Group for renal cell carcinoma. Renal cell carcinoma guideline. Eur Urol. 2007 Jun;51(6):1502-10. doi: 10.1016/j.eururo.2007.03.035. Epub 2007 Mar 28. PMID 17408850
- [Result] Cheng C, Lu M, Zhang Y, Hu X. Effect of augmented reality navigation technology on perioperative safety in partial nephrectomies: A meta-analysis and systematic review. Front Surg. 2023 Apr 12;10:1067275. doi: 10.3389/fsurg.2023.1067275. eCollection 2023. PMID 37123539
- [Result] Thompson RH, Lane BR, Lohse CM, Leibovich BC, Fergany A, Frank I, Gill IS, Blute ML, Campbell SC. Renal function after partial nephrectomy: effect of warm ischemia relative to quantity and quality of preserved kidney. Urology. 2012 Feb;79(2):356-60. doi: 10.1016/j.urology.2011.10.031. PMID 22310752
- [Result] Desai MM, de Castro Abreu AL, Leslie S, Cai J, Huang EY, Lewandowski PM, Lee D, Dharmaraja A, Berger AK, Goh A, Ukimura O, Aron M, Gill IS. Robotic partial nephrectomy with superselective versus main artery clamping: a retrospective comparison. Eur Urol. 2014 Oct;66(4):713-9. doi: 10.1016/j.eururo.2014.01.017. Epub 2014 Jan 25. PMID 24486306
- [Result] Piramide F, Kowalewski KF, Cacciamani G, Rivero Belenchon I, Taratkin M, Carbonara U, Marchioni M, De Groote R, Knipper S, Pecoraro A, Turri F, Dell'Oglio P, Puliatti S, Amparore D, Volpi G, Campi R, Larcher A, Mottrie A, Breda A, Minervini A, Ghazi A, Dasgupta P, Gozen A, Autorino R, Fiori C, Di Dio M, Gomez Rivas J, Porpiglia F, Checcucci E; European Association of Urology Young Academic Urologists and the European Section of Uro-Technology. Three-dimensional Model-assisted Minimally Invasive Partial Nephrectomy: A Systematic Review with Meta-analysis of Comparative Studies. Eur Urol Oncol. 2022 Dec;5(6):640-650. doi: 10.1016/j.euo.2022.09.003. Epub 2022 Oct 7. PMID 36216739
- [Result] Mir MC, Ercole C, Takagi T, Zhang Z, Velet L, Remer EM, Demirjian S, Campbell SC. Decline in renal function after partial nephrectomy: etiology and prevention. J Urol. 2015 Jun;193(6):1889-98. doi: 10.1016/j.juro.2015.01.093. Epub 2015 Jan 29. PMID 25637858
- [Result] Minervini A, Carini M. Tumor Enucleation Is Appropriate During Partial Nephrectomy. Eur Urol Focus. 2019 Nov;5(6):923-924. doi: 10.1016/j.euf.2019.02.009. Epub 2019 Feb 21. PMID 30797738
- [Result] Yu J, Xie HUA, Wang S. The effectiveness of augmented reality assisted technology on LPN: a systematic review and meta-analysis. Minim Invasive Ther Allied Technol. 2022 Oct;31(7):981-991. doi: 10.1080/13645706.2022.2051190. Epub 2022 Mar 25. PMID 35337249
- [Result] Wang J, Lu Y, Wu G, Wang T, Wang Y, Zhao H, Zhou Z, Wu J. The role of three-dimensional reconstruction in laparoscopic partial nephrectomy for complex renal tumors. World J Surg Oncol. 2019 Sep 11;17(1):159. doi: 10.1186/s12957-019-1701-x. PMID 31511081
- [Result] Di Maida F, Campi R, Lane BR, De Cobelli O, Sanguedolce F, Hatzichristodoulou G, Antonelli A, Grosso AA, Noyes S, Rodriguez-Faba O, Keeley FX, Langenhuijsen J, Musi G, Klatte T, Roscigno M, Akdogan B, Furlan M, Simeone C, Karakoyunlu N, Marszalek M, Capitanio U, Volpe A, Brookman-May S, Gschwend JE, Smaldone MC, Uzzo RG, Kutikov A, Minervini A, Sib International Consortium. Predictors of Positive Surgical Margins after Robot-Assisted Partial Nephrectomy for Localized Renal Tumors: Insights from a Large Multicenter International Prospective Observational Project (The Surface-Intermediate-Base Margin Score Consortium). J Clin Med. 2022 Mar 23;11(7):1765. doi: 10.3390/jcm11071765. PMID 35407375
- [Result] Alaraimi B, El Bakbak W, Sarker S, Makkiyah S, Al-Marzouq A, Goriparthi R, Bouhelal A, Quan V, Patel B. A randomized prospective study comparing acquisition of laparoscopic skills in three-dimensional (3D) vs. two-dimensional (2D) laparoscopy. World J Surg. 2014 Nov;38(11):2746-52. doi: 10.1007/s00268-014-2674-0. PMID 25002241
- [Result] Vettoretto N, Foglia E, Ferrario L, Arezzo A, Cirocchi R, Cocorullo G, Curro G, Marchi D, Portale G, Gerardi C, Nocco U, Tringali M, Anania G, Piccoli M, Silecchia G, Morino M, Valeri A, Lettieri E. Why laparoscopists may opt for three-dimensional view: a summary of the full HTA report on 3D versus 2D laparoscopy by S.I.C.E. (Societa Italiana di Chirurgia Endoscopica e Nuove Tecnologie). Surg Endosc. 2018 Jun;32(6):2986-2993. doi: 10.1007/s00464-017-6006-y. Epub 2018 Jan 24. PMID 29368286
- [Result] Checcucci E, Amparore D, Fiori C, Manfredi M, Ivano M, Di Dio M, Niculescu G, Piramide F, Cattaneo G, Piazzolla P, Cacciamani GE, Autorino R, Porpiglia F. 3D imaging applications for robotic urologic surgery: an ESUT YAUWP review. World J Urol. 2020 Apr;38(4):869-881. doi: 10.1007/s00345-019-02922-4. Epub 2019 Aug 27. PMID 31456017